CLINICAL TRIAL: NCT00224718
Title: ACE Trial :Not Worn-Out Aneurism of the Abdominal Aorta Under Renal " Surgery Versus Endoprosthesis "
Brief Title: Elective Abdominal Aortic Aneurism - Open Versus Endovascular Repair
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cecile Jourdain / Project manager, Departement Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P000708; AOM 98167
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-02

CONDITIONS: Elective Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm; Endograft; Open repair; Endovascular repair; AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): surgery - open repair
  Interventions: Procedure: Open repair
- 2 (Experimental): endovascular procedure
  Interventions: Procedure: Endovascular repair (with endograft)

INTERVENTIONS:
Procedure: Endovascular repair (with endograft) — An endovascular stent graft is a tube composed of fabric supported by a metal mesh called a stent. It can be used for a variety of conditions involving the blood vessels, but most commonly to reinforce a weak spot in an artery called an aneurysm. Over time, blood pressure and other factors can cause this weak area to bulge like a balloon and eventually enlarge and rupture. The stent graft seals tightly with your artery above and below the aneurysm. The graft is stronger than the weakened artery and allows blood to pass through it without pushing on the bulge. Physicians typically use endovascular stent grafting to treat abdominal aortic aneurysms (AAAs).
  Arms: 2
Procedure: Open repair — Conventional repair consist in open repair. Different types of surgery can be done : minimal incision aortic surgery (MIAS), transperitoneal approach (TPA), retroperitoneal repair, or conventional median laparotomy.
  Arms: 1

SUMMARY:
Abdominal aortic aneurysm (AAA) is a life threatening disease. There is a consensus to propose surgical repair in patients with a reasonable operative risk when the AAA exceeds 5 cm in diameter.

The aim of the study is to compare the mortality and the occurrence of severe general, vascular and local complications in two groups of patients treated by either by open surgery or by EVAR (EndoVascular Aneurysm Repair). The main outcome criteria and the secondary endpoint are respectively the survival without severe complications and minor morbidity.

DETAILED DESCRIPTION:
ACE Trial :Not Worn-Out Aneurism of the Abdominal Aorta Under Renal " Surgery Versus Endoprosthesis Abdominal aortic aneurysm (AAA) is a life threatening disease. There is a consensus to propose surgical repair in patients with a reasonable operative risk when the AAA exceeds 5 cm in diameter.

The aim of the study is to compare the mortality and the occurrence of severe general, vascular and local complications in two groups of patients treated by either by open surgery or by EVAR (EndoVascular Aneurysm Repair). The main outcome criteria and the secondary endpoint are respectively the survival without severe complications and minor morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years old or more (more than 80 possible depending on physiological age)
* Level 0, 1, or 2 of operative risk
* Abdominal aortic aneurysm with a diameter > or equal to 50 mm or > or equal to 40 mm if rapid growing (10 mm or more in a year), or painful, or saccular aneurysms, or aneurisms of common iliac arteries with a diameter equal or superior to 30 mm; or women with a diameter equal to 45 mm;
* Aortic neck superior or equal to 1.5 cm
* No stenosis superior or equal to 75% of the superior mesenteric artery
* Proximal neck angulation inferior to 80°
* Diameter of the iliac arteries compatible with introducer sheath
* Inform consent signed

Exclusion Criteria:

* Aneurysm involving the renal arteries or with the length of the neck less than 1.5 cm
* Thrombus or major calcification in the neck
* Diameter of the iliac arteries not compatible with introducer sheath
* Level 3 of operative risk
* History of major iodine allergy (Quincke oedema, anaphylactic shock)
* Other comorbidity with life expectancy less than 6 months
* Follow up impossible during the trial
* Participation in another trial
* Inform consent not signed

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2003-01; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Death and major adverse events | 4 years

SECONDARY OUTCOMES:
Minor adverse events (systemic vascular or non vascular complications) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Yann JOUSSET, MD, Principal Investigator — CHU Angers - Hôtel Dieu; Jean M Pernes, MD, Principal Investigator — Hôpital privé d'Antony; Pierre Y Meaulle, MD, Principal Investigator — Clinique mutualiste des Eaux Claires, Grenoble; Jean P Favre, MD, Principal Investigator — CHU Hôpital Nord, Saint-Etienne; Jacques Watelet, MD, Principal Investigator — Hôpital Charles Nicolle, Rouen; Patrick Lermusiaux, MD, Principal Investigator — CHRU -Hôpital Trousseau, Tours; Jean F Heautot, MD, Principal Investigator — CHU de Pontchaillou, Rennes; Mohamad KOUSSA, MD, Principal Investigator — Hôpital Cardiologique , Lille; Patrice BERGERON, MD, Principal Investigator — Hôpital St Joseph, Marseille; Philippe CHAILLOU, MD, Principal Investigator — Hôpital Nord Laennec, Nantes; Eric CHEYSSON, MD, Principal Investigator — Centre Hospitalier René Dubos, Pontoise; Arnaud DEMON, MD, Principal Investigator — CH de Valenciennes; Jean C PILLET, MD, Principal Investigator — Nouvelles Cliniques Nantaises, Nantes; Eric STEINMETZ, MD, Principal Investigator — CHU de Dijon - Hôpital du Bocage; Michel LEVADE, MD, Principal Investigator — Clinique Pasteur Toulouse; Jean CARDON, MD, Principal Investigator — Clinique des Franciscaines, Nimes; Pierre-Edouard MAGNAN, MD, Principal Investigator — CHU Timone, Marseille; Michel Batt, MD, Principal Investigator — Hôpital St-Roch, Nice; Pierre GOUNY, MD, Principal Investigator — Hopital de la cavale blanche, Brest; Antoine Lucas, MD, Principal Investigator — CHU Pontchaillou; Jean P Becquemin, MD, Study Chair — Hopital Henri Mondor, Créteil; Marc Sapoval, MD, Study Chair — HEGP, Paris
Locations (1):
- Hopital Henri Mondor, Créteil, France

REFERENCES:
- [Background] Lederle FA. Endovascular repair of abdominal aortic aneurysm--round two. N Engl J Med. 2005 Jun 9;352(23):2443-5. doi: 10.1056/NEJMe058126. No abstract available. PMID 15944430
- [Derived] Becquemin JP, Pillet JC, Lescalie F, Sapoval M, Goueffic Y, Lermusiaux P, Steinmetz E, Marzelle J; ACE trialists. A randomized controlled trial of endovascular aneurysm repair versus open surgery for abdominal aortic aneurysms in low- to moderate-risk patients. J Vasc Surg. 2011 May;53(5):1167-1173.e1. doi: 10.1016/j.jvs.2010.10.124. Epub 2011 Jan 26. PMID 21276681
- See also: controversies and updates in vascular surgery — http://www.cacvs.org